CLINICAL TRIAL: NCT00719420
Title: A Randomized Clinical Trial to Examine the Efficacy of a Clarithromycin-, Amoxicillin-, and Metronidazole-Based Regimen to Eradicate Helicobacter Pylori Infections in Pasto, Colombia
Brief Title: Clarithromycin, Amoxicillin, and Metronidazole Based Regimens to Treat Helicobacter Pylori Infections in Colombia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of North Texas Health Science Center (Other)
Collaborators: Universidad del Valle, Colombia (Other); Vanderbilt University (Other)
Responsible Party: Dr. Lori A. Fischbach, University of North Texas Health Science Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06-02-24-2
Record Dates: First submitted 2008-07-11; First posted 2008-07-21 (Estimated); Last update posted 2008-07-21 (Estimated); Status verified 2008-07

CONDITIONS: Helicobacter Pylori Infection
Keywords: Randomized clinical trial; Helicobacter pylori; clarithromycin; metronidazole; amoxicillin; proton pump inhibitor; Colombia
MeSH Terms: interventions — Clarithromycin; Metronidazole; Amoxicillin; Omeprazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Clarithromycin 500 mg bid, metronidazole 500 mg tid, and amoxicillin 500mg tid for 14 days (with or without omeprazole 20 mg bid)
  Interventions: Drug: Clarithromycin, Metronidazole, Amoxicillin (+Omeprazole)
- 2 (Active Comparator): Clarithromycin 500 mg bid, amoxicillin 1 g bid, and omeprazole 20 mg bid for 10 days
  Interventions: Drug: Clarithromycin, Amoxicillin, Omeprazole

INTERVENTIONS:
Drug: Clarithromycin, Metronidazole, Amoxicillin (+Omeprazole) — Clarithromycin 500 mg bid, metronidazole 500 mg tid, and amoxicillin 500mg tid with or without omeprazole 20 mg bid for 14 days
  Other Names: Biaxin, Flagyl, Amoxil, Prilosec
  Arms: 1
Drug: Clarithromycin, Amoxicillin, Omeprazole — Clarithromycin 500 mg bid, amoxicillin 1 g bid, and omeprazole 20 mg bid for 10 days
  Other Names: Biaxin, Amoxil, Prilosec
  Arms: 2

SUMMARY:
More than half of the world's population is infected with Helicobacter pylori, a bacterium that colonizes the human stomach. Although most infected subjects live free of symptoms and disease outcomes (except superficial gastritis), only a few develop peptic ulcers or gastric cancer, while some others may develop non-ulcer dyspepsia. Current clinical practice for the management of peptic ulcer disease includes testing for and treating H. pylori, if present. Although there are triple therapies that contain 2 antibiotics plus a bismuth compound, a proton-pump inhibitor, or a H2-receptor antagonist which are effective at eliminating H. pylori in Europe and North America, these treatments are dramatically less effective in developing countries. Our recent meta-analysis showed quadruple therapies containing clarithromycin, amoxicillin, metronidazole and a proton pump inhibitor to be effective in the presence of clarithromycin or metronidazole resistance. However, this regimen has yet to be tested in a developing country. Therefore, in the current randomized clinical trial in Pasto, Colombia, we aim to examine the effectiveness of clarithromycin, amoxicillin, metronidazole with and without a proton pump inhibitor compared to the Food and Drug Administration approved 10-day regimen containing clarithromycin, amoxicillin and omeprazole. Since antibiotic therapy is most effective within a specific gastric pH range, and since mutifocal atrophy results in damage and loss of the acid producing parietal cells, we will test the efficacy of our modified therapy stratified by diagnosis of multifocal atrophic gastritis.

DETAILED DESCRIPTION:
Warren and Marshall's Noble prize winning discovery of Helicobacter pylori, and their subsequent work which showed that gastritis and peptic ulcers could be successfully treated by eradicating this bacterium, ultimately revolutionized how physicians treat peptic ulcer disease. However, our previous research has shown most treatments for H. pylori are dramatically less effective in the presence of drug resistance, especially in developing countries, where H. pylori is highly prevalent. Our recent meta-analysis, which prompted the Canadian Helicobacter Consensus Group to change their treatment guidelines for Canada, showed quadruple therapies of clarithromycin, amoxicillin, metronidazole (CAM) and a proton pump inhibitor to be effective in the presence of clarithromycin or metronidazole resistance. However, this regimen has yet to be tested in a developing country.

Since Warren and Marshall's discovery, H pylori has also been implicated as a risk factor for gastric cancer and possibly non-ulcer dyspepsia (NUD), while conflicting evidence suggests it may be a protective factor for disease outcomes of the esophagus. Glandular atrophy caused by H. pylori is believed to initiate the precancerous process by disrupting the mucus barrier, allowing carcinogens direct contact to gastric cells. Atrophy is followed by an increase in pH in the gastric cavity. Carcinogens, epithelium mutations, rapid cell turnover, toxins, and virulence factors such as H. pylori strains containing CagA and vacuolating cytotoxin (VacA) proteins, and the cagA and vacA genes that encode for these proteins, are putative risk factors for progression to intestinal metaplasia, followed by dysplasia, and then invasive carcinoma.

Much debate exists about whether anti H. pylori treatments benefit infected subjects with non-ulcer dyspepsia. A meta-analysis of short-term trials suggest that H. pylori is a weak risk factor for dyspepsia in some unidentified populations. This information together with a cost-effectiveness analysis resulted in the European Maastricht 2-2000 Consensus recommendation that young patients with persistent dyspepsia be tested and, if infected, treated for H. pylori ('the test-and-treat strategy'). Nevertheless, without strong evidence supporting this strategy for dyspepsia, and devoid of an understanding of how H. pylori elimination affects symptoms, this strategy has not gained wide spread acceptance and it is not part of the current standard of care in many countries. However, studies which examine the effect of H. pylori on symptoms in developing countries, where most infections occur, are lacking.

Although gastric cancer rates have declined in developed countries, higher rates have been observed in minority and immigrant groups, and it is still the 2nd most frequent cancer worldwide. In Nariño, Colombia, the incidence for gastric cancer is estimated to be the highest in the world with a rate up to 150/100,000/yr. In 1993-94 we conducted a randomized clinical trial aimed at short-term reduction of inflammation and epithelial damage in the stomachs of H. pylori infected subjects with NUD from the general population of Pasto, the capital of Nariño (the "Pasto cohort"). Data from this trial and our subsequent meta-analysis showed that classical anti-H. pylori treatments which effectively eliminate H. pylori in Europe and North America, were not effective in populations such as Pasto which has a high prevalence of the infection and a high prevalence of metronidazole resistance.

We will test the efficacy of promising 14-day clarithromycin-, amoxicillin- and metronidazole-(CAM) triple and quadruple based regimens for eradication compared with the FDA recommended 10-day regimen (clarithromycin, amoxicillin, and omeprazole). Since antibiotic therapy is most effective within a specific gastric pH range, and since mutifocal atrophy results in damage and loss of the acid producing parietal cells, we will test the efficacy of our modified therapy stratified by diagnosis of multifocal atrophic gastritis. We hypothesize that: 1) among H. pylori infected subjects in the Pasto cohort with multifocal atrophic gastritis, those who are randomized to a 14-day triple therapy with CAM will more likely eradicate their H. pylori infection compared with those randomized to the FDA approved regimen; 2) among H. pylori infected subjects in the Pasto cohort without multifocal atrophic gastritis, those who are randomized to a 14-day quadruple therapy of CAM plus omeprazole, will be more likely eradicate their H. pylori infection compared with those randomized to the FDA approved regimen; and 3) among H. pylori infected subjects in Pasto without a previous histological diagnosis, those randomized to a 14-day CAM therapy will be more likely to eradicate H. pylori compared with those randomized to the FDA approved regimen. Therefore, our primary aim is to conduct a randomized clinical trial in Pasto, Colombia to assess the diagnosis-specific efficacy of a 14-day CAM triple therapy, and a 14-day clarithromycin, amoxicillin, metronidazole and omeprazole quadruple therapy to eliminate H. pylori compared with the FDA approved 10-day clarithromycin, amoxicillin, and omeprazole triple therapy in subjects who have never been treated for H pylori infection.

ELIGIBILITY:
Inclusion Criteria:

* Aged 29-77 years; have lived in Pasto, Colombia for at least 5 years and plan to remain in Pasto for ≥5 more years;
* Currently have Helicobacter pylori infection;
* Willing to refrain from alcohol consumption for 2 weeks;
* Have never taken a therapy to eradicate Helicobacter pylori;
* Have not taken antibiotics, bismuth compounds, proton-pump inhibitors, H2-receptor antagonists, or antacids within 30 days of the trial;
* Are not pregnant, and have little or no risk of pregnancy.

Exclusion Criteria:

* History of kidney, liver, heart, or mental disease;
* Frequent alcohol consumption;
* Allergic to clarithromycin, amoxicillin, penicillin, omeprazole or metronidazole;
* Currently taking drugs which may interact with any of the trial medications.

Ages: 29 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2006-04; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Helicobacter pylori eradication determined by 13C-urea breath test. | 4-6 weeks following the completion of treatment

SECONDARY OUTCOMES:
Dyspeptic symptom resolution ascertained by self-report. | 4-6 weeks following the completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Lori A Fischbach, PhD, MPH, Principal Investigator — University of North Texas Health Science Center; Pelayo Correa, MD, Study Chair — Vanderbilt University; Luis E Bravo, MD, Study Director — Universidad del Valle
Locations (1):
- Universidad del Valle, Cali, Colombia

REFERENCES:
- [Derived] Fischbach LA, Bravo LE, Zarama GR, Bravo JC, Ojha RP, Priest EL, Collazos T, Casabon AL, Guerrero LZ, Singh KP, Correa P. A randomized clinical trial to determine the efficacy of regimens containing clarithromycin, metronidazole, and amoxicillin among histologic subgroups for Helicobacter pylori eradication in a developing country. Helicobacter. 2009 Apr;14(2):100-8. doi: 10.1111/j.1523-5378.2009.00667.x. PMID 19298337